CLINICAL TRIAL: NCT06730035
Title: PRediction of Outcomes and PERsonalized Radiotherapy by Biomarkers and Functional Imaging
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROPER; Ricerca Corrente 2022-2024 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2024-12-01; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Rectal Cancer, Radiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental analysis on tissues (Experimental): The results obtained from the study should not be considered conclusive but rather as generators of research hypotheses for potential subsequent studies to be conducted on larger populations.
  Interventions: Other: Blood analysis

INTERVENTIONS:
Other: Blood analysis — This is an experimental analysis on tissues (peripheral blood) and exploratory, which is why the enrollment of a limited number of patients has been planned. The results obtained from the study should not be considered conclusive but rather as generators of research hypotheses for potential subsequent studies to be conducted on larger populations. The qualitative and quantitative characteristics of the vesicles and their miRNA content will be analyzed descriptively.

SUMMARY:
This is a study focused on analyses of peripheral blood (tissue study). The aim of the trial is to determine whether it is possible to predict early clinical and/or pathological responses after radiotherapy in the setting of neoadjuvant treatment for locally advanced rectal carcinomas, through qualitative and quantitative assessment of circulating extracellular vesicles in plasma and the microRNA (miRNA) contained within them. Extracellular vesicles are "clean-up" structures that collect various elements circulating in the blood, including fragments of DNA and RNA from tumor cells. Observing how these structures and their contents change with radiotherapy could provide early indications of the tumor's response to treatment. The trial seeks to answer the question: "Can the quantity of CD69+ vesicles in patients undergoing neoadjuvant radiotherapy predict their response early?"

The trial is monocentric and plans to enroll approximately 30 patients. Participation in this trial does not offer direct benefits, as it involves only laboratory investigations without modifications to the usual diagnostic-therapeutic process for the condition considered.

The collection of information is aimed at improving knowledge regarding extracellular vesicles. These vesicles could provide early insights into the response to neoadjuvant radiotherapy for locally advanced rectal tumors. In this way, subsequent therapeutic strategies can be personalized based on this response.

DETAILED DESCRIPTION:
This is a monocentric, exploratory experimental study on tissues (peripheral blood), which is why the enrollment of a limited number of patients has been planned. The results obtained from the study should not be considered conclusive but rather as generators of research hypotheses for potential subsequent studies to be conducted on larger populations. The qualitative and quantitative characteristics of the vesicles and their miRNA content will be analyzed descriptively.

The primary objective will be considered achieved if values of CD69+ vesicles > 349 absolute units correctly predict the response to radiotherapy in at least 80% of patients. Subsequently, the investigators aim to verify if CD86+ vesicles > 10 absolute units and CD3+ > 4 absolute units correctly predict the response to radiotherapy in at least 80% of cases. Additionally, the association between the values of the three indicated vesicles (both original and dichotomized as above or below the specified cut-offs, derived from preliminary results of our research group) and the time to disease recurrence at two years will be tested.

Patients will be treated according to clinical practice in accordance with the physician's judgment and the information provided in the Technical Data Sheet of each individual product of any concomitant therapies administered as per clinical practice. The diagnostic-therapeutic pathway of the patients will not be influenced in any way by the results of tissue tests conducted for the study.

The TC-PET investigations, as part of the normal diagnostic-therapeutic process, will be performed at the Nuclear Medicine Unit of the IRCCS University Hospital of Bologna. Molecular investigations will be carried out at the laboratory of the Immunogenetics and Transplant Biology Unit (IBT) affiliated with the IRCCS University Hospital of Bologna, S. Orsola Polyclinic. The study is aimed at patients undergoing neoadjuvant RT for locally advanced rectal tumors within one year. The study is expected to begin on 01/05/2023, and in any case, only after approval from the Ethics Committee and the subsequent release of the company's authorization.

Patients will be enrolled during the first visit at the Radiotherapy Unit of the IRCCS University Hospital of Bologna, prior to any sampling necessary for the specific study analyses. It should be noted that investigations on the total quantification of DNA and epigenetic changes (methylation and miRNA expression) do not involve genome sequencing. The DNA molecules will be examined without considering individual specificity; therefore, the individual's genetic code remains unknown after the examination. A sample of 10 ml of venous blood will be collected using a vacutainer with EDTA from each patient, and plasma will be collected for each experimental point. Biological samples will be pseudonymized and labeled with the progressive number RT/NEO/00N. All samples will be stored in specially marked RT containers in a locked freezer located in the IBT laboratory until their use. Transport will be carried out using a sealed and temperature-controlled dedicated container by the personnel involved in the project.

Three samples will be analyzed per patient: 1st sample: 1-5 days before the start of RT, 2nd sample: at the end of the 3rd week of RT, 3rd sample: on the last day of RT. Therefore, a total of 90 samples are expected to be analyzed.

Isolation of Nanovesicles: plasma samples will be processed for the separation of extracellular vesicles through column gel ultrafiltration with sterilized and buffered CL-B4 resin. The nanovesicles will then be processed for phenotypic analysis using the Miltenyi MACSPEX kit and processed for DNA/RNA extraction using the Nucleo Spin Tissue kit (Macherey Nagel, M-Medical, Milan, Italy). The procedure will be carried out at the IBT laboratory of the IRCCS University Hospital of Bologna.

Epigenetic Analysis:

* MicroRNA Analysis The RNA samples extracted from the extracellular vesicles will be analyzed for microRNA content using Droplet Digital PCR at the IBT laboratory.
* Methylation Analysis The DNA methylation profile analysis of nucleated blood cells will be conducted using mass spectrometry performed on the Sequenom platform and the EpiTyper protocol (Sequenom) at the IBT laboratory of the IRCCS University Hospital of Bologna. All statistical analyses will be performed at the IBT unit.

Visits, assessments, and systemic and local treatments will be carried out according to clinical practice and will not be altered for this study. The aliquots of peripheral blood required for the specific study analyses will be collected in addition to routine samples taken during patient treatments and follow-ups, using the same venous access. Specifically, the samples will be taken at the start of radiotherapy, three weeks after the start, and at the end, within the context of exams and visits scheduled by normal clinical practice.

During the first visit, according to clinical practice, information related to the patient's clinical history (oncological history, remote pathological history, pharmacological history, family history) will be collected. A general physical examination will be performed, and the radiotherapy pathway will be planned. The patient's eligibility for the PROPER study will be assessed, and if affirmative, informed consents will be obtained.

Analysis Methodology:

The demographic and clinical characteristics of the patients will be described using median and interquartile range (for continuous variables) and absolute frequencies and percentages (for categorical variables).

The evaluation of the predictive capability of the vesicles will be performed through sensitivity and specificity analysis of the predefined cutoffs (CD69+ > 349 absolute units; CD86+ > 10 absolute units; CD3+ > 4 absolute units) to verify that all have a positive predictive value (PPV) > 80%. ROC analysis using the original values of the vesicles will also be conducted to identify any alternative cutoff values that may better discriminate regarding the outcome.

The analysis of disease-free survival at two years from the start of therapy will be conducted descriptively using Kaplan-Meier curves and the log-rank test. Patients who died due to fatal complications will be censored at the date of death. Given the small size of the study population, Cox regressions may be performed, including the indicator of whether the vesicular cutoff was exceeded as a risk factor, along with a maximum of one confounder, provided that the number of events (disease recurrences) is adequate for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients candidates for neoadjuvant RT, administered with hypofractionated-accelerated treatment, for locally advanced rectal tumors;
* Age ≥ 18 years
* Obtaining informed consent

Exclusion Criteria:

* Contraindications to MRI, uncontrolled chronic intestinal diseases or pelvic infections
* Pregnancy and breastfeeding
* Unwillingness to participate in follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Pathological response | through study completion, an average of 1 year
  The response to therapy will be assessed as a complete pathological response, defined as present/absent according to the staging criteria commonly used in clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Giuseppe Morganti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Italy